CLINICAL TRIAL: NCT05504447
Title: To Evaluate the Efficacy and Safety of "Rongyang Zhengyifang" Tea Bag in Mildly Diagnosed Patients With COVID-19 Variant Virus
Brief Title: To Evaluate the Efficacy and Safety of "Rongyang Zhengyifang" Tea Bag With COVID-19 Variant Virus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2022-06-007B
Record Dates: First submitted 2022-08-16; First posted 2022-08-17 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Herbal Interaction

STUDY DESIGN:
Intervention Model Description: 1. Parallel study design.
  2. There is a control group (placebo).
  3. Blinding method: non-blind.
  4. Random assignment: yes
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rong-Yang Zhengyifang" tea bag (Experimental): 1. Inclusion criteria:
     Aged over 20 years old, according to the guidelines of the Epidemic Command Center, during home isolation and self-epidemic prevention or home quarantine, use a household novel coronavirus antigen rapid screening reagent to test positive, and after the medical staff confirms the relevant symptoms or the PCR test is positive, it is determined to be mild. Those who were diagnosed with severe disease and who did not use antiviral drugs were given tea immediately.
  2. Exclusion criteria:
  (1)Patient characteristics: excluded under 20 years of age, incapacity, pregnancy or lactation women (2)Disease characteristics: Western medicine has clearly diagnosed mental diseases (3)Environmental characteristics: Other conditions that prevent the patient from cooperating. If you feel unwell after screening not to sign the subject's consent form, etc.
  Interventions: Other: Rong-Yang Zhengyifang" tea bag
- placebo tea bag (Placebo Comparator): The appearance is exactly the same as the Zhengyifang tea bag, and the ingredient is oolong tea
  Interventions: Other: placebo tea bag

INTERVENTIONS:
Other: Rong-Yang Zhengyifang" tea bag — One tea bag is 4 grams, 3 bags per day, for a total of 7 days
  Arms: Rong-Yang Zhengyifang" tea bag
Other: placebo tea bag — One tea bag is 4 grams, 3 bags per day, for a total of 7 days
  Arms: placebo tea bag

SUMMARY:
The strategy of our study is to use traditional Chinese medicine tea to regulate physical fitness and strength can be enhanced to help patients with mildly diagnosed COVID-19 variant virus to achieve self-recovery ability and avoid the development of moderate and severe symptoms.

DETAILED DESCRIPTION:
According to the "Interim Guidelines for the Clinical Treatment of Novel Coronavirus SARS-CoV-2 Infection" published by the CDC of the Ministry of Health and Welfare on June 23, 2021, it can be classified into mild, moderate, severe and extremely severe according to the classification of its related clinical manifestations.

Current clinical studies have found that COVID-19 primarily attacks the bronchioles and alveoli of the lower respiratory tract. In severe cases, it may induce an inflammatory response, leading to pulmonary airway and alveolar damage, and even pulmonary fibrosis.

The strategy of our study is to use traditional Chinese medicine tea to regulate physical fitness and strength can be enhanced to help patients with mildly diagnosed COVID-19 variant virus to achieve self-recovery ability and avoid the development of moderate and severe symptoms.It may reduce the expenditure of health insurance and medical expenses, and more importantly, if it can be administered timely to block the progression of the disease when mild-to-moderate symptoms occur, it can also reduce the burden of hospital medical care.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 20 years old, according to the guidelines of the Epidemic Command Center, during home isolation and self-epidemic prevention or home quarantine period, use the home novel coronavirus antigen rapid screening reagent to test positive, and after the medical staff confirms the relevant symptoms or the PCR test is positive, it is determined as Those who were mildly diagnosed and who did not use antiviral drugs were given tea immediately.

Exclusion Criteria:

* Patient characteristics: Exclude women under the age of 20, incapacitated, pregnant or breastfeeding
* Disease characteristics: subjects who have been diagnosed with mental illness by Western medicine, and who have long-term diarrhea or long-term use of traditional Chinese medicine
* Environmental characteristics: other conditions that prevent the patient from cooperating. Such as being unsuitable after screening, not signing the subject's consent form, etc.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Questionnaire Evaluation | 7days
  The questionnaire contains a total of 28 assessment items:
  Divided into 7 major aspects: nasal symptoms (6 questions), eye symptoms (2 questions), Sleep condition (4 questions), ear symptoms (5 questions), overall symptoms (7 questions), daily life Influence (4 questions) and the influence of emotions (3 questions). According to the patient's 7 days,the symptoms within are scored for each item, and the first category is to evaluate the symptoms of this item. The first score ranges from 0 points (no such symptoms) to 5 points (extremely severe Heavy); The second category is to assess the importance of this symptom to the patient, starting from 1 Points (not important) to 4 points (very important). Multiply these two fractions together to get the symptom-impact score , this is the individual evaluation score of each patient for each symptom.

SECONDARY OUTCOMES:
Rapid screening reagent screening | 7days
  Comparison of the number of days from a positive diagnosis of rapid screening to a negative test

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Ying Kung, doctor, Study Chair — TaipeiVGH Center for Traditional Medicine
Locations (1):
- Center for Traditional Medicine, Taipei Veterans General Hospital, Taipei County, Taiwan